CLINICAL TRIAL: NCT04934878
Title: Regional Treatment Flow and Prognosis ofTraumatic Thoracic Aortic Injuries：A Multi-center Retrospective Analysis in Zhejiang Province During 11 Years
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hwa Mei Hospital, University of Chinese Academy of Sciences (Unknown); Zhoushan Hospital Zhejiang Province (Unknown); Taizhou Hospital Zhejiang Province (Unknown); Quzhou People's Hospital Zhejiang Province (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Shaoxing People's Hospital (Other); Ningbo No. 1 Hospital (Other); The Central Hospital of Lishui City (Other); Ningbo Medical Center Li Huili Hospital (Unknown); Lishui People's Medical (Unknown); Jinhua Central Hospital (Other); 903 Hospital of Chinese People's Liberation Army (Other); Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other); First People's Hospital of Hangzhou (Other); Zhejiang Quhua Hospital (Other); Yinzhou Second Hospital (Unknown); Tiantai County People's Hospital (Unknown); Taizhou Hospital (Other); The First People's Hospital of Huzhou (Other); Suichang County People's Hospital (Unknown); Quzhou Second People's Hospital (Unknown); Ningbo Fenghua District People's Hospital (Unknown); Jiangshan People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-859
Record Dates: First submitted 2021-06-05; First posted 2021-06-22 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-05

CONDITIONS: Severe Trauma; Blunt Thoracic Aortic Injury; Interventional Therapy; Treatment Protocal
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Referral information: first visit to our hospital/transfer from another hospital
  Interventions: Biological: Referral information

INTERVENTIONS:
Biological: Referral information — first visit to our hospital/transfer from another hospital

SUMMARY:
Using keywords (main) artery dissection aneurysm (main) artery haematoma (main) To diagnose X-ray imaging reports and medical record home page is a search, check the unit 11 hospitals in Zhejiang Province during the year aortic injury clinical data of 11 years, through the electronic questionnaire to fill in the form of information, information of diagnosis and treatment of the basic information for the patient injury mechanism and so on carries on the statistical analysis. Basic information includes gender, age, history of hypertension. Injury information includes injury mechanism information and trauma information. Injury mechanism refers to injuries caused by car accidents, high falls and other causes. Injury information includes diagnosis, injury severity score, Glasgow coma index, and Stanford classification of aortic injury. The information of diagnosis and treatment includes the method of treatment, the reason for referral, the time of definitive treatment and the prognosis. The method of treatment is divided into the first treatment group and the referral group. The first treatment group refers to the patients admitted by the hospital for the first time, and the referral group refers to the patients transferred from other hospitals. The reasons for referral include: the suggestion of the hospital after comprehensive consideration, the lack of diagnosis and treatment qualification of the hospital, the subjective will of the patient's family members. Deterministic treatment time refers to the time from injury to imaging examination and the time from injury to surgery and other data to be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of trauma patients with aortic dissection (aortic aneurysm) (aortic hematoma)

Exclusion Criteria:

* Patients with primary aortic dissection, limb pseudoaneurysm, non-aortic associated hematoma, etc.Incomplete or lost data, patients refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Regional Treatment Flow And Prognosis of Traumatic Thoracic Aortic Injuries：A Multi-Center Retrospective Analysis in Zhejiang Province During 11 Years | From January 2010 to October 2020,
  Numbers of hospitals of different levels
Regional Treatment Flow And Prognosis of Traumatic Thoracic Aortic Injuries：A Multi-Center Retrospective Analysis in Zhejiang Province During 11 Years | From January 2010 to October 2020,
  Number of Stanford type(A and B)
Regional Treatment Flow And Prognosis of Traumatic Thoracic Aortic Injuries：A Multi-Center Retrospective Analysis in Zhejiang Province During 11 Years | From January 2010 to October 2020,
  survial rate

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZU, Hanzhou, Zhejiang, China